CLINICAL TRIAL: NCT00558012
Title: Maintenance of Skeletal Integrity in Frail Elders
Brief Title: Zoledronic Acid for Osteoporosis in the Elderly
Acronym: ZEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0612018; R01AG028086-01A1 (NIH)
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Osteoporosis; Bone Loss; Fragility Fractures
Keywords: Osteoporosis; Bone loss; Frail Geriatric Women; Nursing Home Patients; Fragility Fractures
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Zoledronic Acid; Vitamin D; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Medication Group (Experimental): One-time dose: Intravenous Zoledronic Acid 5.0 mg; Vitamin D (800 IU/daily); Calcium 1200 mg/daily (supplement plus diet)
  Interventions: Drug: Intravenous zoledronic acid; Dietary Supplement: Vitamin D 800 IU/daily; Dietary Supplement: Calcium 1200 mg/daily
- Placebo (Placebo Comparator): One-time dose: intravenous saline; Vitamin D (800 IU/daily); 1200 mg calcium (supplement plus diet)
  Interventions: Drug: Intravenous zoledronic acid; Dietary Supplement: Vitamin D 800 IU/daily; Dietary Supplement: Calcium 1200 mg/daily

INTERVENTIONS:
Drug: Intravenous zoledronic acid — Intravenous zoledronic acid 5.0 mg once
  Other Names: Zometa; Reclast
Dietary Supplement: Vitamin D 800 IU/daily — Daily divided dose
Dietary Supplement: Calcium 1200 mg/daily — supplement plus diet

SUMMARY:
This trial will examine the safety, efficacy and feasibility of a single dose of intravenous zoledronic acid in the maintenance of skeletal integrity for frail, institutionalized women, who are most at risk for the deleterious outcomes of osteoporosis. The investigators will test the hypothesis that in institutionalized elderly women a single dose of intravenous zoledronic acid therapy will: (1) be efficacious as demonstrated by stability or improvement in bone mass measurements and reductions in bone turnover; (2) be safe and feasible; and (3) provide estimates for vertebral and nonvertebral fracture reduction in this cohort for use in planning a future study.

DETAILED DESCRIPTION:
This is a 2-year, randomized, double-blind, calcium/vitamin D-controlled clinical trial of a single dose of therapy with at least 12 months follow-up. All participants will receive calcium and vitamin D throughout the trial. At baseline, 190 women will be randomized in a 1:1 allocation to zoledronic acid (group 1) or zoledronic acid placebo (group 2). At the end of 24 months, women will be followed to gather data on longer term fragility fracture rates and survival until all participants have completed 24 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* We will include elderly women 65 years and older if they reside in a nursing home or an assisted living facility and have a known history of osteoporosis, as determined by history of an adult fragility fracture or bone mineral density criteria for osteoporosis (T-score -2.5 at the total hip, femoral neck or spine) or low bone mass (T-score < -2.0 at the total hip, femoral neck or spine, consistent with the National Osteoporosis Foundation Treatment guidelines). If a participant's spine and or hip are not evaluable (due to surgery, calcifications, artifact in the scan area, scoliosis, etc.), they may be included in the study with a T-score of ≤ -2.0 at the forearm.
* Elders will be chosen without consideration of ethnic or racial background. We chose frail, institutionalized women because 70-85% of them have osteoporosis and this age group is substantially under-treated.
* We will include all who qualify, if they are able to weight bear or assist with transfer to chair, to endure that the results have maximum generalizability to the nursing home population as a whole.

Exclusion Criteria:

* Children will be excluded because they are not frail, institutionalized elders.
* Men will be excluded because they do not become postmenopausal and are less likely to become osteoporotic.
* We will exclude institutionalized women with subacute illnesses who are not expected to survive or who will be discharged in less than 2 years.
* We will also exclude patient with a contraindication to bisphosphonate, such as hypocalcemia, allergy, pervious adverse event (excluding gastrointestinal disorders), or currently on an oral bisphosphonate.
* We will exclude patients with a calculated creatinine clearance of < 30 ml/mm.
* We will exclude women scheduled for or in need of a tooth extraction as this procedure has been associated with osteonecrosis of the jaw in patients with cancer given multiple coursed of high dose intravenous bisphosphonates.
* We will screen for these conditions by detailed history, physical exam (including dental exam), chart review, and baseline laboratory analyses, including BUN/creatinine, liver function tests, TSH, calcium, PTH, 25-hydroxyvitamin D, alkaline phosphatase and baseline calculated creatinine clearance. Participants with vitamin D levels < 20 ng/ml will be treated with vitamin D 50,000 IU/wk for 8 weeks in addition to calcium. Vitamin D will be rechecked and the patient will be enrolled if the vitamin D level is > 20 ng/ml.
* Patients will be allowed to continue on certain medications known to affect bone and mineral metabolism (e.g. glucocorticoids, anticonvulsants) because their use is common in this population. (In our facilities, 2.9% of patients use glucocorticoids and 7.2% use anti-epileptic drugs.) In addition, women who have been treated in the past or present with osteoporosis agents, such as estrogen/progesterone, raloxifene, and calcitonin, will be allowed to participate and continue on these therapies if prescribed by their physician. However, if patients are currently on or have been on bisphosphonates for greater than 1 year in the previous 2 years prior to enrollment, they will be excluded as some bisphosphonates are long acting.
* Patients will be allowed to wear hip pads if prescribed by their physician. If they are on parathyroid hormone, they may participate, but will be told that monotherapy with parathyroid hormone is more beneficial than combination therapy with parathyroid hormone and alendronate, as we have previously demonstrated.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 181 (Actual)
Dates: Start 2007-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Greenspan SL, Perera S, Ferchak MA, Nace DA, Resnick NM. Efficacy and safety of single-dose zoledronic acid for osteoporosis in frail elderly women: a randomized clinical trial. JAMA Intern Med. 2015 Jun;175(6):913-21. doi: 10.1001/jamainternmed.2015.0747. PMID 25867538

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Medication Group: One-time dose: Intravenous Zoledronic Acid 5.0 mg
  Intravenous zoledronic acid: Intravenous zoledronic acid 5.0 mg once
- Placebo: Placebo
  One-time dose: Intravenous saline
Period: Overall Study
Arm/Group | Active Medication Group | Placebo
Started | 89 | 92
Completed | 64 | 74
Not Completed | 25 | 18

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo
  Intravenous zoledronic acid: Intravenous zoledronic acid 5.0 mg once
- Total: Total of all reporting groups
Arm/Group | Active Medication Group | Placebo | Total
Number analyzed (Participants) | 89 | 92 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 89 | 92 | 181
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 92 | 181
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 89 | 92 | 181

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD) of the Total Hip and Spine
Description: BMD is the bone mineral density of the lumbar spine and total hip measured using dual-energy xray absorptiometry (DXA) scan
Time Frame: Baseline, 12 months, 24 month
Population: Number of patients that completed a DXA at 12 months. At 24 months 60 in active treatment group and 72 in placebo group completed a DXA.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Active Medication Group | Placebo
Number analyzed (Participants) | 75 | 83
Percent change
  Spine BMD at 24 months | 4.5 (0.8) | 0.7 (0.5)
  Spine BMD at 12 months | 3.0 (0.5) | 1.1 (0.5)
  Total Hip BMD at 24 months | 2.6 (0.6) | -1.5 (0.7)
  Total Hip BMD at 12 months | 2.8 (0.5) | -0.5 (0.4)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Active Medication Group | Placebo
Serious Adverse Events (participants affected / at risk) | 60/89 | 55/92
Other Adverse Events (participants affected / at risk) | 87/89 | 88/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Medication Group (N=89) | Placebo (N=92)
Atrial fibrillation (Cardiac disorders) | 3 | 3
choroid melanoma (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 8 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 4 | 1
Arterial bypass operation (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 6 | 3
Chest pain (Cardiac disorders) | 1 | 7
Myocardial infarction (Cardiac disorders) | 2 | 1
Oedema perepheral (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Clostridium difficile colitis (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Diverticulitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastoenteritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Gastriesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Proctitis ulcerative (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 5
Fall (Injury, poisoning and procedural complications) | 4 | 4
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Post traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Sepsis (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Femur fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Fractured sacrum (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pubic rami fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Tibia fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Confusional state (Nervous system disorders) | 1 | 0
Dementia Alzheimers type (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 3 | 2
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 3 | 4
Tremor (Nervous system disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 4 | 4
Urosepsis (Renal and urinary disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Knee arthroplast (Surgical and medical procedures) | 1 | 2
Shoulder arthroplasty (Surgical and medical procedures) | 0 | 2
Arteriosclerosis (Vascular disorders) | 0 | 2
Colitis ischaemic (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Labile blood pressure (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Medication Group (N=89) | Placebo (N=92)
Atrial fibrillation (Cardiac disorders) | 5 | 5
Diarrhea (Gastrointestinal disorders) | 7 | 12
Death (General disorders) | 8 | 3
Bronchitis (Infections and infestations) | 6 | 3
Contusion (Injury, poisoning and procedural complications) | 5 | 13
Anorexia (Metabolism and nutrition disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 7
Headache (Nervous system disorders) | 14 | 8
Urinary tract infection (Renal and urinary disorders) | 16 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Cellulitis (Skin and subcutaneous tissue disorders) | 9 | 7
Tooth extraction (Surgical and medical procedures) | 4 | 5
Ecchymosis (Vascular disorders) | 1 | 5
Cardiac failure congestive (Cardiac disorders) | 8 | 4
Chest pain (Cardiac disorders) | 8 | 12
Oedema peripheral (Cardiac disorders) | 5 | 5
Nausea (Gastrointestinal disorders) | 13 | 7
Fatigue (General disorders) | 24 | 14
Influenza-like illness (General disorders) | 6 | 2
Pyrexia (General disorders) | 8 | 1
Pneumonia (Infections and infestations) | 12 | 9
Fall (Injury, poisoning and procedural complications) | 69 | 54
Infusion site bruising (Injury, poisoning and procedural complications) | 11 | 12
Post traumatic pain (Injury, poisoning and procedural complications) | 5 | 5
Skin laceration (Injury, poisoning and procedural complications) | 8 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 7
Transient ischemic attack (Nervous system disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No